CLINICAL TRIAL: NCT02065531
Title: Effects of Myofascial Soft Tissue Release and Mobilization With Impulse Technique Torsion in Subjects With Chronic Non-specific Low Back Pain: A Randomized Clinical Trial
Brief Title: Myofascial Release and Mobilization With Impulse Technique Torsion in Low Back Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Responsible Party: Principal Investigator, Adelaida María Castro-Sánchez, Lecturer, Universidad de Almeria
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: UAL-021
Record Dates: First submitted 2014-01-10; First posted 2014-02-19 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Low Back Pain; Chronic Disease
Keywords: Low Back Pain; Chronic Pain; Manipulation; Manual Therapy; Randomized Controlled Trial
MeSH Terms: conditions — Low Back Pain; Chronic Disease; Chronic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Myofascial Soft Tissue Release (Experimental): Protocol: Transverse Plane-Level Clavicular Release. Diaphragmatic Transverse Plane Release. Square the Lumbar Fascia Release. Gluteal Fascia Release. Hint Of Pubic Region Release. Fascia Psoas Release. Lumbo-sacral Decompression. Pelvic Floor Release.
  Interventions: Other: Myofascial Soft Tissue Release
- Mobilization with impulse technique (Active Comparator): Subject in lateral decubitus with extension and lower limb traction contact the couch with contralateral lower limb was performed triple flexion and left trunk rotation. This technique reduces the slack (tension joints) of the ventral pelvis, head and into the contralateral side of the sacrum support (base) with the forearm.
  Interventions: Other: Mobilization with impulse technique.

INTERVENTIONS:
Other: Myofascial Soft Tissue Release — Protocol: Transverse Plane-Level Clavicular Release. Diaphragmatic Transverse Plane Release. Square the Lumbar Fascia Release. Gluteal Fascia Release. Hint Of Pubic Region Release. Fascia Psoas Release. Lumbo-sacral Decompression. Pelvic Floor Release.
  Arms: Myofascial Soft Tissue Release
Other: Mobilization with impulse technique. — Subject in lateral decubitus with extension and lower limb traction contact the couch with contralateral lower limb was performed triple flexion and left trunk rotation. This technique reduces the slack (tension joints) of the ventral pelvis, head and into the contralateral side of the sacrum support (base) with the forearm.
  Arms: Mobilization with impulse technique

SUMMARY:
The purpose of the current randomized clinical trial was to compare the effectiveness of myofascial soft tissue release versus mobilization with impulse technique torsion (anterior) on pain, disability, and kinesiophobia in individuals with chronic non-specific low back pain.

DETAILED DESCRIPTION:
Design: Randomized Clinical Trial. Objective: to determine the effects of myofascial soft tissue release versus mobilization with impulse technique torsion (anterior) on pain, disability and kinesiophobia in individuals with chronic non-specific low back pain.

Methods and Measures: sixty-four individuals will be randomly assigned to one of two groups.

Intervention: For 12-week, the group 1 will undergo treatment comprising a myofascial soft tissue release protocol (1/week) and the group 2 will receive a mobilization with impulse technique torsion (anterior) (1/week).

Main Outcome Measures: Intensity of pain, disability, fear of movement, isometric endurance of trunk flexor muscles and lumbar mobility in flexion data will be collected at baseline, and 24hr after the last manual therapy application. Mixed-model analyses of variance will be used to examine the effects of the treatment on each outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Score ≥4 on the Roland Morris Disability Questionnaire
* Inability to achieve lumbar muscle flexion-relaxation in trunk flexion
* Low back pain for ≥3 months
* Not undergoing another physical therapy treatment

Exclusion Criteria:

* Disease of the central or peripheral nervous system
* Having previously undergone spinal manipulative therapy
* Contraindication to low back thrust manipulation
* A history of spinal surgery
* Treatment with corticosteroid in the past two weeks
* Clinical signs of radiculopathy
* Presence of lumbar stenosis
* Diagnosis of spondylolisthesis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Roland Morris Disability Questionnaire (RMDQ) | At baseline, 12 weeks and 16 weeks
  This is a self-reported questionnaire consisting of 24 items reflecting limitations in different activities of daily living attributed to low back pain including walking, bending over, sitting, lying down, dressing, sleeping, self-care and daily activities.

SECONDARY OUTCOMES:
Change from baseline in Oswestry Low Back Pain Disability Index (ODI) | At baseline, 12 weeks and 16 weeks
  The ODI has 10 items referring to activities of daily living that might be disrupted by low back pain. Each item is answered on a 6-point Likert scale ranging from "no problem at all" [0] to "not possible" [5]. The total score ranges from 0 to 50.
Change from baseline in Numerical Pain Rating Scale | At baseline, 12 weeks and 16 weeks
  A 10-point Numerical Pain Rating Scale (NPRS; 0: no pain, 10: maximum pain) assesses the patients' current level of pain, and the worst and lowest level of pain experienced in the preceding 24 hours.
Change from baseline in Tampa Scale of Kinesiophobia | At baseline, 12 weeks and 16 weeks
  The Tampa Scale of Kinesiophobia (TSK) is a 17-item questionnaire developed to measure the fear of movement and (re)injury. Each item is scored on a four-point Likert scale ranging from "strongly disagree" [1] to "strongly agree" [4].
Change from baseline in Isometric endurance of trunk flexor muscles | At baseline, 12 weeks and 16 weeks
  The McQuade test measures the isometric resistance of abdominal muscles in seconds.
Change from baseline in Lumbar mobility in flexion | At baseline, 12 weeks and 16 weeks
  Lumbar mobility in flexion is determined by measuring the finger-to-floor distance with a tape.

CONTACTS AND LOCATIONS:
Overall Officials: Adelaida Castro-Sánchez, Lecturer, Principal Investigator — Universidad de Almeria
Locations (1):
- Universidad de Almeria, Almería, Almería, Spain

REFERENCES:
- [Background] Cymet TC. Osteopathic manual treatment and ultrasound therapy for chronic low back pain: an illustration of osteopathic semantic confusion. J Am Osteopath Assoc. 2014 Jan;114(1):6-7. doi: 10.7556/jaoa.2014.002. No abstract available. PMID 24384968
- [Background] Hidalgo B, Hall T, Nielens H, Detrembleur C. Intertester agreement and validity of identifying lumbar pain provocative movement patterns using active and passive accessory movement tests. J Manipulative Physiol Ther. 2014 Feb;37(2):105-15. doi: 10.1016/j.jmpt.2013.09.006. Epub 2014 Jan 6. PMID 24401656
- [Background] Ebert R, Campbell A, Kemp-Smith K, O'Sullivan P. Lumbar spine side bending is reduced in end range extension compared to neutral and end range flexion postures. Man Ther. 2014 Apr;19(2):114-8. doi: 10.1016/j.math.2013.08.004. Epub 2013 Sep 4. PMID 24315299
- [Background] Rabin A, Shashua A, Pizem K, Dickstein R, Dar G. A clinical prediction rule to identify patients with low back pain who are likely to experience short-term success following lumbar stabilization exercises: a randomized controlled validation study. J Orthop Sports Phys Ther. 2014 Jan;44(1):6-B13. doi: 10.2519/jospt.2014.4888. Epub 2013 Nov 21. PMID 24261926
- [Background] Zimney K, Louw A, Puentedura EJ. Use of Therapeutic Neuroscience Education to address psychosocial factors associated with acute low back pain: a case report. Physiother Theory Pract. 2014 Apr;30(3):202-9. doi: 10.3109/09593985.2013.856508. Epub 2013 Nov 19. PMID 24252071
- [Background] Haskins R, Osmotherly PG, Southgate E, Rivett DA. Physiotherapists' knowledge, attitudes and practices regarding clinical prediction rules for low back pain. Man Ther. 2014 Apr;19(2):142-51. doi: 10.1016/j.math.2013.09.005. Epub 2013 Oct 3. PMID 24176916
- [Background] Licciardone JC. Osteopathic manual treatment and ultrasound therapy for chronic low back pain: an illustration of osteopathic semantic confusion. Author reply. J Am Osteopath Assoc. 2013 Sep;113(9):661-2. doi: 10.7556/jaoa.2013.031. No abstract available. PMID 24133757
- [Background] Kumar S, Beaton K, Hughes T. The effectiveness of massage therapy for the treatment of nonspecific low back pain: a systematic review of systematic reviews. Int J Gen Med. 2013 Sep 4;6:733-41. doi: 10.2147/IJGM.S50243. PMID 24043951
- [Background] Leysen P, Bombeke K, Remmen R. Osteopathic manual treatment and ultrasound therapy for chronic low back pain: an illustration of osteopathic semantic confusion. J Am Osteopath Assoc. 2013 Sep;113(9):660-1. doi: 10.7556/jaoa.2013.030. No abstract available. PMID 24005084
- [Background] Bachmann S, Oesch P. [Physiotherapy and rehabilitation for low back pain]. Ther Umsch. 2013 Sep;70(9):543-8. doi: 10.1024/0040-5930/a000444. German. PMID 23985153
- [Background] Hands-on treatment helps low back pain. Harv Womens Health Watch. 2013 Jun;20(10):8. No abstract available. PMID 23977709
- [Background] Eirikstoft H, Kongsted A. Patient characteristics in low back pain subgroups based on an existing classification system. A descriptive cohort study in chiropractic practice. Man Ther. 2014 Feb;19(1):65-71. doi: 10.1016/j.math.2013.07.007. Epub 2013 Aug 6. PMID 23932099
- [Background] Muir JM. Chiropractic management of a patient with low back pain and Castellvi type II lumbosacral transitional vertebrae. J Chiropr Med. 2012 Dec;11(4):254-9. doi: 10.1016/j.jcm.2012.02.005. PMID 23843757
- [Background] Donaldson M, Learman K, O'Halloran B, Showalter C, Cook C. The role of patients' expectation of appropriate initial manual therapy treatment in outcomes for patients with low back pain. J Manipulative Physiol Ther. 2013 Jun;36(5):276-83. doi: 10.1016/j.jmpt.2013.05.016. PMID 23829882